CLINICAL TRIAL: NCT02991092
Title: The Influence of Different Fluid Therapy Measures on the Postoperative Outcome in Fast Track of Colon Cancer After Laparoscopic Surgery.
Brief Title: The Influence of Different Fluid Therapy Measures on the Postoperative Outcome in Fast Track of Colon Cancer.（FTSlapCC)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Quan Wang (Other)
Responsible Party: Sponsor-Investigator, Quan Wang, Deputy chief physician, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FTSlapCC
Record Dates: First submitted 2016-11-30; First posted 2016-12-13 (Estimated); Last update posted 2016-12-13 (Estimated); Status verified 2016-12

CONDITIONS: Colon Carcinoma
Keywords: colon carcinoma; liquid treatment; fast-track surgery
MeSH Terms: conditions — Colonic Neoplasms | interventions — Hypodermoclysis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- the experimental group (Experimental): After surgery, patients in the experiment group were provided with intravenous fluid administration at 1.0ml/Kg/h and encouraged to take food and drink water early after surgery, and the intravenous fluid administration was stopped immediately when the oral intake was more than 1500ml/h
  Interventions: Procedure: fluid administration
- the control group (Other): patients in the control group strictly followed the fasting and were provided with the intravenous fluid administration according to "Total amount of fluid = physiological requirement + additional loss (fever + gastrointestinal decompression) + amount lost" until their intestinal function completely recovered.
  Interventions: Procedure: fluid administration

INTERVENTIONS:
Procedure: fluid administration — After surgery, patients in the experiment group were provided with intravenous fluid administration at 1.0ml/Kg/h and encouraged to take food and drink water early after surgery, and the intravenous fluid administration was stopped immediately when the oral intake was more than 1500ml/h; patients in the control group strictly followed the fasting and were provided with the intravenous fluid administration according to "Total amount of fluid = physiological requirement + additional loss (fever + gastrointestinal decompression) + amount lost" until their intestinal function completely recovered.

SUMMARY:
To compare the influence of two different fluid administration strategies on the clinical efficacy of patients with colorectal carcinoma during the fast-track surgery.

DETAILED DESCRIPTION:
Patients that were diagnosed with colorectal carcinoma by the First Hospital of Jilin University and were scheduled to undergo the laparoscopic surgery were prospectively included and divided into the experimental group and the control group with the random number method. After surgery, patients in the experiment group were provided with intravenous fluid administration at 1.0ml/Kg/h and encouraged to take food and drink water early after surgery, and the intravenous fluid administration was stopped immediately when the oral intake was more than 1500ml/h; patients in the control group strictly followed the fasting and were provided with the intravenous fluid administration according to "Total amount of fluid = physiological requirement + additional loss (fever + gastrointestinal decompression) + amount lost" until their intestinal function completely recovered. The blood volume change indicators (heart rate, mean arterial pressure, oxyhemoglobin saturation, inferior vena cava diameter /body surface area (VCD), intra-abdominal pressure, specific gravity of urine, BNP, etc.) and inflammation indicators (CRP, IL-6, TNF-a) of the two groups of patients were observed and a comparison was made of the recovery time of intestinal function, incidence of complications, hospitalization time after operation and hospitalization expenses of the two groups.

ELIGIBILITY:
Inclusion Criteria:

1. the age of 18-70 years old
2. the pathological diagnosis of colon cancer patients
3. no surgical intervention.

Exclusion Criteria:

1. patients with heart, lung, liver, renal function were significantly abnormal
2. body mass index kg >35 / m2
3. pregnancy
4. sepsis or systemic inflammatory response syndrome patients.
5. patients with severe malnutrition.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-11; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
recovery time of intestinal function | within the first 30 days (plus or minus 3 days) after surgery

SECONDARY OUTCOMES:
TNF-alpha | the first day to the forth day After the operation
CRP[=C reactive protein]ba | the first day to the forth day After the operation
IL-10[=interleukin-10] | the first day to the forth day After the operation
BNP[=type B natriuretic peptide] | the first day to the forth day After the operation
hospitalization time after operation（day） | within the first 30 days (plus or minus 3 days) after surgery

OTHER OUTCOMES:
inferior vena cava diameter（mm） | Twenty-fourth hours after operation and before operation
stat body height（m） | Twenty-fourth hours after operation and before operation
body weight（Kg） | Twenty-fourth hours after operation and before operation

CONTACTS AND LOCATIONS:
Overall Officials: Shengk Qiu, master, Principal Investigator — qiusk7009@sina.com

IPD SHARING:
Plan to Share IPD: Undecided